CLINICAL TRIAL: NCT02811510
Title: Gender Related Differences in the Acute Effects of Delta-9-Tetrahydrocannabinol in Healthy Humans: Sub-Study I
Acronym: THC-Gender-I
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mohini Ranganathan, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1505015940.A
Record Dates: First submitted 2016-06-02; First posted 2016-06-23 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- THC (Active Comparator): 10 mg Dronabinol will be administered orally.
  Interventions: Drug: Dronabinol
- Placebo (Placebo Comparator): Placebo pill (no active cannabinoids).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo pill (no active cannabinoids)
  Arms: Placebo
Drug: Dronabinol — 10 mg capsule of Dronabinol will be administered orally.
  Other Names: Delta-9-Tetrahydrocannabinol
  Arms: THC

SUMMARY:
The purpose of the study is to characterize the acute effects of cannabinoids in women relative to men and to begin probing the mechanisms that may underlie gender differences.

DETAILED DESCRIPTION:
To characterize the acute effects of oral Dronabinol (10 mg capsule) in women relative to men and to begin probing the mechanisms that may underlie gender differences.

ELIGIBILITY:
Inclusion Criteria:

* At least one lifetime exposure to cannabis
* Good physical and mental health

Exclusion Criteria:

* Cannabis naive individuals
* Major current or recent stressors
* Taking estrogen supplements or oral contraceptive pills (for women)
* Sesame oil allergy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline: Rewarding Effects measured by Visual Analog Scale (VAS) | changes in "high" assessed over the following timepoints: baseline, +60, +80, +120, +180, +300 minutes after start of oral Dronabinol administration.
  Subjective measure of THC induced "high"
Change from Baseline: Verbal Learning: Measured by Rey Auditory Verbal Learning Test (RAVLT) | baseline and +80 minutes after start of oral Dronabinol administration.
  Measured as delay recall on the AVLT

CONTACTS AND LOCATIONS:
Locations (1):
- Biological Studies Unit at the VA Connecticut Healthcare System, Yale School of Medicine, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No